CLINICAL TRIAL: NCT01724138
Title: An Open Label Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Efficacy of Deferasirox Administered to Chinese Patients With β-thalassemia Major Aged From 2 to Less Than 6 Years Old
Acronym: MACS2163
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670ACN02
Record Dates: First submitted 2012-10-24; First posted 2012-11-09 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2014-08

CONDITIONS: β-thalassemia Major
Keywords: deferasirox
MeSH Terms: interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferasirox (Experimental): The study will provide PK, safety, tolerability and efficacy data collected during 48 weeks of treatment with deferasirox in Chinese pediatric patients with transfusion dependent -thalassemia major, aged 2 to <6 years at enrollment. The target patient pool consists of 20 patients with evidence of iron overload measured by serum ferritin level at the start of study. Patients will start their deferasirox treatment with a dose of 20 mg/kg/day. Serum ferritin will be monitored every month and the dose of deferasirox will be adjusted if necessary every 3 months based on the trends in serum ferritin. Other possible dose adjustments will be based on the patient's safety assessments.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Patients will start their deferasirox treatment with a dose of 20 mg/kg/day.

SUMMARY:
To characterize the PK of deferasirox in pediatric β-thalassemia major patients aged from 2 to less than 6 years old, when administrated with a fixed starting dose of 20 mg/kg/day.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged from 2 to less than 6 years old.
* Patients with transfusion dependent β-thalassemia major.
* Serum ferritin values ≥ 1000 ng/ml at screening.
* Written informed consent must be obtained from the patient's legal guardian in accordance with local law and regulation prior to any screening procedures.

Exclusion Criteria:

* Non-transfusion-dependent thalassemia.
* Systemic diseases which would prevent study treatment (e.g. uncontrolled hypertension, cardiovascular, renal, hepatic, metabolic, etc.)
* Serum creatinine > age adjusted ULN.
* Significant proteinuria as indicated by a urinary protein/creatinine ratio (UPCR) ≥ 0.5mg/mg in a non-first void urine sample at screening. If UPCR is found to be ≥ 0.5 mg/mg the test can be repeated after 1 month.
* ALT/AST > 2.5xULN and total bilirubin > 1×ULN.
* Left ventricular ejection fraction < 56% by echocardiography.
* Patient has a known history of HIV seropositivity or history of active/treated hepatitis B or C (a test for screening is not required).
* A history of clinically relevant ocular and/or auditory toxicity related to iron chelation therapy
* Any surgical or medical conditions which will significantly alter the absorption, distribution, metabolism or excretion of the drug(e.g. ulcerative disease, uncontrolled nausea, vomiting, malabsorption syndrome, obstruction, or stomach and/or small bowel resection).
* Other conditions which investigator deems potential harm to patients if participate the study.

Ages: 2 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
the PK profile of deferasirox in pediatric β-thalassemia major patients aged from 2 to less than 6 years old. | PK sampling times are 0.5, 2.5, 6, 10h in Day 1 postdose; Day 2, 3, 4 and 5 predose and 0.5, 2.5, 6, 10h post dose on Day 4, then pre-dose at each subsequent visit until Week 49. Day -1 PK sample will be treated as Day 1 predose sample.
  Area under the plasma concentration-time curve from time zero to the end of the dosing interval.
the PK profile of deferasirox in pediatric β-thalassemia major patients aged from 2 to less than 6 years old: Cmax | PK sampling times are 0.5, 2.5, 6, 10h in Day 1 postdose; Day 2, 3, 4 and 5 predose and 0.5, 2.5, 6, 10h post dose on Day 4, then pre-dose at each subsequent visit until Week 49. Day -1 PK sample will be treated as Day 1 predose sample.
  The maximum plasma concentration of study medication.
the PK profile of deferasirox in pediatric β-thalassemia major patients aged from 2 to less than 6 years old: Tmax | PK sampling times are 0.5, 2.5, 6, 10h in Day 1 postdose; Day 2, 3, 4 and 5 predose and 0.5, 2.5, 6, 10h post dose on Day 4, then pre-dose at each subsequent visit until Week 49. Day -1 PK sample will be treated as Day 1 predose sample.
  Tmax was directly determined from the raw plasma concentration-time data.

SECONDARY OUTCOMES:
The safety and tolerability of deferasirox following multiple dosing in pediatric β-thalassemia major patients. | Baseline, every 4 weeks until 48 weeks after taking the drug
  The adverse events and abnormal measurements of hematology, blood chemistry, urinalysis, urinary protein/creatinine ratio, physical examination, auditory and ocular examinations, ECG, ECHO, and growth development are collected for the measurement of safety and tolerability.
The efficacy of deferasirox in pediatric β-thalassemia patients as measured by change of serum ferritin. | Baseline, every 4 weeks until 48 weeks after taking the drug
  Changes in serum ferritin from baseline to every 4 weeks are collected for the measurement of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals